CLINICAL TRIAL: NCT00817180
Title: Multi-centre, Long-term Comparative Trial of High Frequency Chest Wall Oscillation Versus Positive Expiratory Pressure Mask in the Treatment of Cystic Fibrosis
Brief Title: Long-term Study, Comparing Vest Therapy to Positive Expiratory Pressure (PEP) Therapy in the Treatment of Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H07-03181; CW08-0128
Record Dates: First submitted 2009-01-02; First posted 2009-01-06 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Cystic Fibrosis
Keywords: physiotherapy; airway clearance techniques; Positive Expiratory Pressure Technique; high frequency Chest Wall Oscillation; vest
MeSH Terms: conditions — Cystic Fibrosis | interventions — Positive-Pressure Respiration; Chest Wall Oscillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Positive Expiratory Pressure (PEP) - an airway clearance technique
  Interventions: Other: Positive Expiratory Pressure (PEP)
- B (Active Comparator): High Frequency Chest Wall Oscillation (HFCWO) also known as the 'Vest technique' - an airway clearance technique.
  Interventions: Other: High Frequency Chest Wall Oscillation (HFCWO) using InCourage Vest System

INTERVENTIONS:
Other: Positive Expiratory Pressure (PEP) — Physiotherapy technique for airway clearance
  Arms: A
Other: High Frequency Chest Wall Oscillation (HFCWO) using InCourage Vest System — Physiotherapy technique for airway clearance.
  Arms: B

SUMMARY:
This study is a preliminary study designed to determine the safety and effectiveness of HFCWO using the InCourage vest system as an airway clearance technique for the treatment of CF. The study will compare HFCWO to the most commonly used airway clearance technique in Canada, namely the Positive Expiratory Pressure technique in patients with CF over a period of one year. As this is a preliminary study, it will not be able to determine if the vest is equivelant to PEP, but will provide the information needed to plan a larger study to answer that question.

DETAILED DESCRIPTION:
Objective This is a pilot study to evaluate the long-term clinical efficacy of high frequency chest wall oscillation (HFCWO) using the inCourage vest system, compared to positive expiratory pressure mask (PEP) in the treatment of patients with cystic fibrosis.

Study Design This is a one year prospective multi-centre randomized controlled trial of HFCWO versus PEP as airway clearance techniques in patients with cystic fibrosis. Number of respiratory exacerbations will be compared between the two treatment arms. Slope of percent predicted in FEV1, activity level, quality of life, cost analysis and subject satisfaction will also be compared.

Number of subjects Enrollment will be completed after 170 subjects have been recruited, approximately 85 in each arm.

Number of sites The study will involve between 14 CF centres in Canada.

PERSCRIBED AIRWAY CLEARANCE TECHNIQUE The test airway clearance technique is the

* High Frequency Chest Wall Oscillation using the InCourage Vest System. This will be compared to
* The Positive Expiratory Pressure Mask Technique. Subjects will be randomized to perform one of these techniques as their airway clearance technique for the period of the study.

PRIMARY ENDPOINT Primary: Difference in the number of respiratory exacerbations. (For definition see Appendix A). Defined by the presence of one major criteria or 2 minor signs or symptoms.

Major Criteria:

* Decrease in FEV1 of ≥10% from best baseline within past 6 months, unresponsive to ventolin.
* Oxygen saturation <90% on room air or ≥ 5% decline from previous baseline.
* New finding(s) on chest radiograph.
* Hemoptysis (more than streaks on more than one occasion in past week).

Minor Signs/symptoms:

* Increased work of breathing or respiratory rate.
* New or increased adventitial sounds on lung exam.
* Weight loss ≥ 5% of body weight or decrease across one major percentile in weight percentile for age within the past 6 months.
* Increased cough.
* Decreased exercise tolerance or level of activity.
* Increased chest congestion or change in sputum.

For minor signs/symptoms, duration of symptoms need to be ≥ 5 days or significant symptom severity.

SECONDARY ENDPOINTS

Secondary:

* The time to the first respiratory exacerbation will be measured in each group using the same definition of a respiratory exacerbation as used for the primary outcome.
* Change in FEV1 measured as difference in the yearly mean rate of decline (Appendix E).
* Cost analysis between the two groups.
* Quality of life questionnaire.
* Patient satisfaction questionnaire.
* Adherence to treatment.

DATA SAFETY MONITORING COMMITTEE

The study will be monitored by a Data Safety Monitoring committee (DSMC). The will communicate regularly either by teleconference, email or by face to face meetings, to deal with issues that arise. The will review all serious adverse events as they occur. The DSMC may request an analysis at any time. At the end of the randomized trial, a report of select final analyses will be provided the DSMC. The study may be terminated if the investigators, medical monitor, or DSMC have significant concerns about the safety of HFCWO based on serious adverse events, other safety data or the conduct of the trial.

STATISTICS Primary Analysis: The number of exacerbations during treatment will be determined in each arm and the difference between the groups calculated with 95% confidence limits as a measure of precision.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 6 years of age or older at enrollment and be competent in performing spirometry.
* Confirmed diagnosis of CF.
* FEV1> 45% predicted as calculated by Wang reference equations
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
* Clinically stable at enrollment with no evidence of respiratory exacerbation within a month of enrollment as assessed by the site CF Physician.
* Willingness to adhere to prescribed treatment regimen.

Exclusion Criteria:

* Diagnosis of Allergic Broncho-Pulmonary Aspergillosis, or a persistent culture for B.cepacia complex within the previous 1 year period
* .On active treatment for non Tuberculous Mycobacterium.
* Use of intravenous antibiotics within the previous 14 days of enrollment.
* Initiation and or change in maintenance therapy within 14 days of enrollment.
* Use of systemic corticosteriods (1mg/kg if < 20 kg or 20 mg of prednisone per day) within 14 days of enrollment.
* Concurrent participation in another study that could potentially affect the present study.
* Haemoptysis of over 20 mls on more than 2 occasions within the previous 30 days from enrollment.
* A pneumothorax in the six months preceding the study.
* Presence of a condition or abnormality that in the opinion of the site CF Physician would compromise the safety of the patient or the quality of the data.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-10; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Difference in the number of respiratory exacerbations during the 1 year study period | 1 year

SECONDARY OUTCOMES:
The time to the first respiratory exacerbation. Change in FEV1 measured as difference in the yearly mean rate of decline. Cost analysis between the two groups. Quality of life questionnaire. Patient satisfaction questionnaire and Adherence to treatment. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Maggie McIlwaine, Physio, Principal Investigator — BC Children's Hospital, Vancouver; George Davidson, MD, Study Director — BC Children's Hospital, Vancouver; Candice Bjornson, MD, Study Director — Alberta Children's Hospital; Clare Smith, Physio, Study Director — Alberta Children's Hospital; Hans Pasterkamp, MD, Study Director — Children's Hospital of Winnipeg; Linda Kraemer, Physio, Study Director — Children's Hospital of Winnipeg; Felix Ratjen, MD, Study Director — The Hospital for Sick Children, Toronto; Jennifer Agnew, Physio, Study Director — The Hospital for Sick Children, Toronto; Larry Lands, MD, Study Director — Montreal Children's Hospital of the MUHC; Nancy Alarie, Physio, Study Director — Montreal Children's Hospital of the MUHC; Pearce Wilcox, MD, Study Director — St. Paul's Hospital, Vancouver; Brigette Wilkins, Physio, Study Director — St. Paul's Hospital, Vancouver; Sherri Katz, MD, Study Director — Children's Hospital of Eastern Ontario, Ottawa; Linda Lapointe, Physio, Study Director — Children's Hospital of Eastern Ontario; Shawn Aaron, MD, Study Director — The Ottawa Hospital; Lynne Orser, Physio, Study Director — The Ottawa Hospital; Harvey Rabin, MD, Study Director — Foothills Medical Centre, Calgary; Julie Wilson, Physio, Study Director — Foothills Medical Centre, Calgary; Mary Noseworthy, MD, Study Director — Janeway Children's Health & Rebab. Centre, St. John's; Stephanie Spencer, Physio, Study Director — St. Clare's Mercy Hospital, St. John's; Peter Zuberbuhler, MD, Study Director — University of Alberta Hospitals, Edmonton; Suzanne Bergsten, Physio, Study Director — University of Alberta Hospitals, Edmonton; Neil Brown, MD, Study Director — University of Alberta Hospitals, Edmonton; Joyce Sharum, Physio, Study Director — University of Alberta Hospitals, Edmonton; Jacques-Edouard Marcotte, MD, Study Director — CHU Ste-Justine, Montreal; Nadia Marquis, Physio, Study Director — CHU Ste-Justine, Montreal; Patrick Daigneault, MD, Study Director — CHUQ, Universite Laval, Quebec; Christine Bouchard, Physio, Study Director — CHUL, Universite Laval, Quebec
Locations (13):
- Canada (13):
  - Foothills Medical Centre, Calgary, Alberta
  - Alberta Children's Hospital, Edmonton, Alberta
  - University of Alberta Hospitals, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Children's Hospital of Winnipeg, Winnipeg, Manitoba
  - St. Clare's Mercy Hospital, St. John's, Newfoundland and Labrador
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - CHU Ste-Justine, Montreal, Quebec
  - Centre Mere-Enfant du CHUQ, Québec, Quebec

REFERENCES:
- [Derived] McIlwaine MP, Alarie N, Davidson GF, Lands LC, Ratjen F, Milner R, Owen B, Agnew JL. Long-term multicentre randomised controlled study of high frequency chest wall oscillation versus positive expiratory pressure mask in cystic fibrosis. Thorax. 2013 Aug;68(8):746-51. doi: 10.1136/thoraxjnl-2012-202915. Epub 2013 Feb 13. PMID 23407019
- See also: Related Info — http://thorax.bmj.com/content/68/8/746.full?sid=cc2c4e5b-3f7c-4edc-9861-b2277ff181bf